CLINICAL TRIAL: NCT02894749
Title: Evaluation of 3D Rotational Angiography After EVAR
Acronym: EVAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departure (and wish not set up study)
Sponsor: University Hospital, Lille (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014_47; 2015-A00645-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Radiation Burn; Aortic Aneurysm, Abdominal
Keywords: hybrid rooms; cone-beam computed tomography
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D Angiography (2DA) (No Intervention): Standard of care - Patients benefit from a 2D completion angiogram at the end of the procedure, and from a angioCT-scan before discharge. If any technical issues is depicted on the CT-scan, a new intervention needs to be scheduled.
- 3D rotational angiography (3DRA) (Experimental): New strategy - Patients benefit from a 3D rotational acquisition at the end of procedure, which offers CT-like reconstructions. If any technical issues is depicted on the 3DRA, it can be treated during the same operating time. A contrast-enhanced ultrasound is performed for each patient before discharge to confirm that no technical issue was missed by the 3DRA.
  Interventions: Radiation: 3D rotational angiography (3DRA)

INTERVENTIONS:
Radiation: 3D rotational angiography (3DRA) — 3DRA allows CT-like reconstructions. It requires less X-rays and contrast medium than standard angioCT-scan. Furthermore, it can be performed in the operative room, during the procedure. Therefore, use of 3DRA should allow reduction of dose, contrast-medium and reintervention when compared to technical success assessment with angioCT-scan.
  Other Names: Cone-beam CT
  Arms: 3D rotational angiography (3DRA)

SUMMARY:
This is a randomized prospective monocentric study to evaluate the benefits of a 3D rotational acquisition (3DRA) to assess technical success after treatment of infra-renal aneurysm with bifurcated endograft. Patients will be randomized between the standard strategy (2D angiography at the end of the procedure and angioCT-scan before discharge) and the new strategy (3DRA at the end of the procedure). Expected findings are a reduction of radiation exposure and contrast medium used during the hospital stay, with a similar resolution between angioCT-scan and 3DRA to depict the main complications after EVAR (occlusion, kinking, endoleak). Furthermore, any complication depicted after 3DRA group could benefit from an additional procedure during the same operating time, and therefore avoid a second intervention for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with EVAR for infra-renal aortic aneurysm
* In a hybrid room
* With a signed consent

Exclusion Criteria:

* Pregnant women
* Patients unable to understand the study protocol or to give their consents
* Renal insufficiency (eGFR<60mL/min)
* Ruptured aneurysms and other emergency settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Effective Dose | Single 1 day - At patient discharge
  Total exposure to radiation in mSv

SECONDARY OUTCOMES:
Contrast Medium | Single 1 day - At patient discharge
  Total amount of contrast medium used (mg of Iodine)
Reintervention rate | During the first 30 days
  Number of secondary procedures due to initial technical issues in both group during the first month
Additional procedure | During surgery
  Number of additional unplanned procedures during the initial operating time, thanks to complications depicted by respectively the 2D angiography or the 3D rotational angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Haulon, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologique, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No